CLINICAL TRIAL: NCT01428180
Title: Changes of Cerebral Tissue Oxygen Saturation During Treatment of Patent Ductus Arteriosus in Neonates
Brief Title: Influence of Treatment for Patent Ductus Arteriosus on Cerebral Oxygenation in Preterm Infants
Status: Completed | Type: Observational
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Manuel Schmid, Dr. med., University of Ulm
Other Study IDs: ULMNEONIRS03
Record Dates: First submitted 2011-08-31; First posted 2011-09-02 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Prematurity of Fetus; Patent Ductus Arteriosus
Keywords: preterm neonates; hemodynamically relevant patent ductus arteriosus
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Indomethacin; Ibuprofen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Indomethacin: Infants treated with Indomethacin
  Interventions: Drug: Indomethacin
- Ibuprofen: Infants treated with Ibuprofen
  Interventions: Drug: Ibuprofen
- Ligation: Infants undergoing surgical ligation
  Interventions: Procedure: Surgical Ligation

INTERVENTIONS:
Drug: Indomethacin — 3 doses of 0,2mg/kg every 12h (first week of life) or every 8h (after first week of life)
  Groups: Indomethacin
Procedure: Surgical Ligation — In nonresponders to medical treatment with persistent hemodynamically relevant patent ductus arteriosus surgical ligation is performed.
  Groups: Ligation
Drug: Ibuprofen — 3 doses every 24h; first dose 10mg/kg, second and third dose 5mg/kg
  Groups: Ibuprofen

SUMMARY:
The purpose of this study is to examine the influence medical or surgical treatment for patent ductus arteriosus in preterm infants on cerebral and renal tissue oxygenation and on cardiac output.

DETAILED DESCRIPTION:
In this observational trial the investigators want to examine whether clinical or echocardiographic parameters of patent ductus arteriosus are related to

* cerebral tissue oxygen saturation, total hemoglobin, fractional tissue oxygen extraction and HbD
* renal tissue oxygen saturation, total hemoglobin, fractional tissue oxygen extraction and HbD

as measured by near infrared spectroscopy

and to

* stroke volume
* cardiac output

as measured by electrical cardiometry.

The investigators want to examine the impact of surgical and medical treatment for patent ductus on these parameters. The investigators want to compare the change of these parameters between responders to medical treatment and nonresponders.

ELIGIBILITY:
Inclusion Criteria:

* Newborn infant below 34 weeks postmenstrual age at the time of birth
* Patent ductus arteriosus with signs of hemodynamic relevance (as judged by the attending neonatologist)
* parental informed consent

Exclusion Criteria:

* Patent ductus arteriosus as part of malformation syndrome
* Additional major cardiovascular malformations

Max Age: 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm neonates with patent ductus arteriosus treated in our hospital
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2011-04; Primary Completion 2012-10 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change of cerebral tissue oxygen saturation during treatment for patent ductus arteriosus | from 10 minutes before start of infusion until 4 hours after end of transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Manuel B Schmid, Dr. med., Principal Investigator — University of Ulm
Locations (1):
- University Medical Center, Ulm, Baden-Wurttemberg, Germany